CLINICAL TRIAL: NCT04578925
Title: Happy, Healthy, Loved: A Mobile-delivered Breastfeeding Self-efficacy Intervention for First Time Parents
Acronym: HHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OhioHealth (Other)
Collaborators: Denison University (Unknown); Claremont McKenna College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1296284
Record Dates: First submitted 2020-07-24; First posted 2020-10-08 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Mother partner pairs will be randomly assigned to the HHL program or care as usual.
Who Masked: Participant
Masking Description: Study staff will randomize patients to the intervention or control arm and not inform subjects of their randomization assignment. Intervention group participants will receive text messages that provide resources and encouragement related to breast-feeding. Control group participants will receive text messages with non-breast-feeding related content.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Happy, Healthy, Loved (Experimental): Both parents will complete surveys on a tablet during the postpartum hospital stay. Surveys cover three topic areas related to breast-feeding; modeling and feedback, partner support, and stress coping. For the next 6 weeks participants' will receive 4 personalized text messages per week based on their tablet survey responses. Participants will be asked one yes/no question each week ("still breastfeeding? Text Y for yes, N for no"). Once a "no" response has been received from a participant, all remaining text messages will emphasize coping and partner support rather than breastfeeding.
  Interventions: Behavioral: Happy, Healthy, Loved
- Control (No Intervention): Control group participants will complete surveys on a tablet during the postpartum hospital stay. Surveys cover three topic areas related to breast-feeding; modeling and feedback, partner support, and stress coping. The control group participants will be sent 4 text messages per week for the first 6 weeks, but the content of the texts will be non-breastfeeding related. The content will instead summarize infant development facts.

INTERVENTIONS:
Behavioral: Happy, Healthy, Loved — A text message based, mobile-device delivered intervention that provides educational information to primiparous mothers and their partners about breast-feeding and coping with stress.
  Arms: Happy, Healthy, Loved

SUMMARY:
The purpose of this study is to test if a mobile device delivered intervention program can improve breast-feeding self-efficacy in primiparous mothers.

DETAILED DESCRIPTION:
The proposed study will test if a mobile device based intervention program, called "Happy, Healthy, Loved (HHL)", will impact breast feeding rates and breastfeeding self-efficacy when compared to care as usual. Primiparous women and their partners will be randomly assigned to the HHL program or usual care.

ELIGIBILITY:
Inclusion Criteria:

1. primiparous mothers,
2. living with a partner or spouse,
3. have an intention to breastfeed their infant for at least 6-weeks postpartum;
4. whose infant is not in the Neonatal Intensive Care Unit,
5. have a mobile phone with text message capability,
6. have no current self-reported depressive episode, and;
7. English as a primary language

Exclusion Criteria:

1. mothers who have other biological children,
2. have infants in the Neonatal Intensive Care Unit,
3. do not have a mobile phone with text message capabilities,
4. report current episodes of depression, or are receiving antidepressant treatment or psychotherapy for depression,
5. have initial study survey that indicates suicide risks (participants who are identified as suicidal ideation at 6 weeks or 6 months will receive further assessment and referral but not be excluded from the program because it may be more harmful and penalizing to remove them from the program if they find it helpful. We will remind the participant that continuing is voluntary and there is no penalty if they wish to discontinue participation)
6. do not speak, read and write English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy: Breastfeeding self-efficacy scale short form | 6 weeks postpartum
  Breastfeeding self-efficacy scale short form (McCarter-Spaulding & Dennis, 2010)- The Breastfeeding self-efficacy scale short form (BSES-SF) will be used to measure breastfeeding self-efficacy. The scores for this scale range from 1-5, with higher scores indicating greater self-efficacy related to breastfeeding.
Breastfeeding Self-Efficacy: Breastfeeding self-efficacy scale short form | 6 months postpartum
  Breastfeeding self-efficacy scale short form (McCarter-Spaulding & Dennis, 2010)- The Breastfeeding self-efficacy scale short form (BSES-SF) will be used to measure breastfeeding self-efficacy. The scores for this scale range from 1-5, with higher scores indicating greater self-efficacy related to breastfeeding.
Breastfeeding Rate | 6 weeks postpartum
  Index of breastfeeding status - Women will be asked to identify the level that accurately described their breastfeeding behaviors within the previous 24 hours. Four levels will be reported: exclusive breastfeeding (breast milk only), partial breastfeeding (breast milk and at least 1 bottle of formula per day), token breastfeeding (breast given to comfort baby not for nutrition), and no breastfeeding. Higher values represent more exclusive breastfeeding.
Breastfeeding Rate | 6 months postpartum
  Index of breastfeeding status - Women will be asked to identify the level that accurately described their breastfeeding behaviors within the previous 24 hours. Four levels will be reported: exclusive breastfeeding (breast milk only), partial breastfeeding (breast milk and at least 1 bottle of formula per day), token breastfeeding (breast given to comfort baby not for nutrition), and no breastfeeding. Higher values represent more exclusive breastfeeding.

SECONDARY OUTCOMES:
Coping Behavior | 6 weeks postpartum
  Brief Coping Orientation to Problems Experienced (COPE) - This 28-item validated scale derived from a previously published measure showing reliability and convergent validity with several established coping measures will be used to identify coping strategies consistent with cognitive-behavioral skills. The scale assesses frequency with which a person uses coping strategies rated on a scale of 1-4. The higher the number indicates a higher frequency.
Coping Behavior | 6 months postpartum
  Brief Coping Orientation to Problems Experienced (COPE) - This 28-item validated scale derived from a previously published measure showing reliability and convergent validity with several established coping measures will be used to identify coping strategies consistent with cognitive-behavioral skills. The scale assesses frequency with which a person uses coping strategies rated on a scale of 1-4. The higher the number indicates a higher frequency.
Postpartum Partner Support | 6 weeks postpartum
  Postpartum Partner Support Scale (PPSS) - The PPSS is a 24-item self-report instrument to assess partner postpartum-specific support. Items are rated on a 4-point Likert-type scale (responses from 1-4) to produce a total score ranging from 24 to 96, with higher scores indicating higher levels of postpartum partner support.
Partner Support | 6 weeks postpartum
  Social Provisions Checklist - This is a 30-item measure of perceived support from the co-parent. The scale covers six provisions of support: guidance, reliable alliance, reassurance of worth, attachment, social integration, and opportunity for nurturance. All items are rated on a 5-point scale for a total score of between 30-120, with higher scores indicating higher levels of support.
Postpartum Partner Support | 6 months postpartum
  Postpartum Partner Support Scale (PPSS) - The PPSS is a 24-item self-report instrument to assess partner postpartum-specific support. Items are rated on a 4-point Likert-type scale (responses from 1-4) to produce a total score ranging from 24 to 96, with higher scores indicating higher levels of postpartum partner support.
Partner Support | 6 months postpartum
  Social Provisions Checklist - This is a 30-item measure of perceived support from the co-parent. The scale covers six provisions of support: guidance, reliable alliance, reassurance of worth, attachment, social integration, and opportunity for nurturance. All items are rated on a 5-point scale for a total score of between 30-120, with higher scores indicating higher levels of support.
Hair Cortisol | 0-2 days postpartum
  A small amount (15-30 mg) of hair from the posterior vertex of the head will be collected. Hair strands will then be cut into 3 cm segments, which based on human scalp hair grows at approximately 1 cm per month, so each of the 3 cm samples will index cortisol output during the three trimesters of pregnancy. If hair is less than 9 cm long, the analysis will include only the number of 3 cm segments available. The wash procedure and steroid extraction will be undertaken using high performance liquid chromatography-mass spectrometry. Additionally, mothers will be asked about their hair histories to use as covariates in analysis along with hair sample. Hair histories include questions related to hair color, salon treatments, sunlight exposure, use of hair products, medications, creams, and hair pieces, style and indoor tanning habits.
Sleep Quality (hair cortisol covariate): Pittsburgh Sleep Quality Index (PSQI) | 0-2 days postpartum
  Pittsburgh Sleep Quality Index (PSQI) - This scale assesses sleep quality, which is a covariate of hair cortisol and mood. The PSQI is well-established questionnaire for assessing sleep quality, duration and disturbances. Items range from 0-3, with high scores indicating greater sleep disturbance.
Postnatal Depression | 0-2 days postpartum
  Edinburgh Postnatal Depression Scale (EPDS) - The EPDS is a well-validated 10-item self-report depression screening tool, in which endorsement of each item is based on how women feel during the previous 7 days. Possible scores range from 0 to 30, with high scores reflecting more depressive symptoms.
Postnatal Depression | 6 weeks postpartum
  Edinburgh Postnatal Depression Scale (EPDS) - The EPDS is a well-validated 10-item self-report depression screening tool, in which endorsement of each item is based on how women feel during the previous 7 days. Possible scores range from 0 to 30, with high scores reflecting more depressive symptoms.
Postnatal Depression | 6 months postpartum
  Edinburgh Postnatal Depression Scale (EPDS) - The EPDS is a well-validated 10-item self-report depression screening tool, in which endorsement of each item is based on how women feel during the previous 7 days. Possible scores range from 0 to 30, with high scores reflecting more depressive symptoms.
Depression, Anxiety, Stress | 0-2 days postpartum
  Depression Anxiety and Stress Scales (DASS-21) - The DASS-21 will be used to measure the unique symptoms of each state. There is normative data for the scale. Scores range from 0-63, with higher scores indicating more severe depression, anxiety, and stress.
Depression, Anxiety, Stress | 6 weeks postpartum
  Depression Anxiety and Stress Scales (DASS-21) - The DASS-21 will be used to measure the unique symptoms of each state. There is normative data for the scale. Scores range from 0-63, with higher scores indicating more severe depression, anxiety, and stress.
Depression, Anxiety, Stress | 6 months postpartum
  Depression Anxiety and Stress Scales (DASS-21) - The DASS-21 will be used to measure the unique symptoms of each state. There is normative data for the scale. Scores range from 0-63, with higher scores indicating more severe depression, anxiety, and stress.
Mood | 0-2 days postpartum
  Maternal Mood Screener (Munoz, 1988) - The mood screener questions were adapted from the Diagnostic Interview Schedule and assesses lifetime and current major depressive episode. Positive endorsement of 5 out of 9 depression symptoms present for at least two weeks screens positive for possible major depressive episode. The screener is a self-report checklist using the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria that has shown high concordance with the Structured Clinical Interview for DSM-IV (SCID-IV), the gold standard diagnostic interview for depression.
Mood | 6 weeks postpartum
  Maternal Mood Screener (Munoz, 1988) - The mood screener questions were adapted from the Diagnostic Interview Schedule and assesses lifetime and current major depressive episode. Positive endorsement of 5 out of 9 depression symptoms present for at least two weeks screens positive for possible major depressive episode. The screener is a self-report checklist using the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria that has shown high concordance with the Structured Clinical Interview for DSM-IV (SCID-IV), the gold standard diagnostic interview for depression.
Mood | 6 months postpartum
  Maternal Mood Screener (Munoz, 1988) - The mood screener questions were adapted from the Diagnostic Interview Schedule and assesses lifetime and current major depressive episode. Positive endorsement of 5 out of 9 depression symptoms present for at least two weeks screens positive for possible major depressive episode. The screener is a self-report checklist using DSM-IV criteria that has shown high concordance with the SCID-IV, the gold standard diagnostic interview for depression.

OTHER OUTCOMES:
Acceptability: Happy Healthy Loved Acceptability Scale | 6 weeks postpartum
  Happy Healthy Loved Acceptability Scale - The investigators developed a list of 11 questions designed to assess participant satisfaction with the program on a scale of 1 (strongly disagree) to 5 (strongly agree). Open ended responses for participants to suggest alterations to the program are included as well.
Acceptability: Happy Healthy Loved Acceptability Scale | 6 months postpartum
  Happy Healthy Loved Acceptability Scale - The investigators developed a list of 11 questions designed to assess participant satisfaction with the program on a scale of 1 (strongly disagree) to 5 (strongly agree). Open ended responses for participants to suggest alterations to the program are included as well.
Adherence | 6 months postpartum
  Adherence will be measured by the percentage of text messages recorded as opened by participants, as well as the percentage of weekly breastfeeding check-in texts participants respond to with a yes, or no response.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Cooper, RN, Principal Investigator — OhioHealth
Locations (1):
- OhioHealth, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Henshaw E, Cooper M, Wood T, Krishna S, Lockhart M, Doan S. A randomized controlled trial of the Happy, Healthy, Loved personalized text-message program for new parent couples: impact on breastfeeding self-efficacy and mood. BMC Pregnancy Childbirth. 2024 Jul 26;24(1):506. doi: 10.1186/s12884-024-06684-9. PMID 39060974

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT04578925/Prot_SAP_002.pdf
  • Informed Consent Form: Maternal Informed Consent (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT04578925/ICF_003.pdf
  • Informed Consent Form: Partner Informed Consent (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT04578925/ICF_004.pdf